CLINICAL TRIAL: NCT05777018
Title: Safety and Efficacy of Ultrasound Guided Lung Recruitment Maneuvers for Prevention of Postoperative Atelectasis After Pediatric Laparoscopic Abdominal Surgery: A Prospective Randomized Study
Brief Title: Ultrasound-guided Lung Recruitment Maneuvers for Postoperative Pediatric Atelectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: atelectasis in pediatrics
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Atelectasis; Postoperative Complications; Recruitment; Pediatric; Abdominal Surgery
MeSH Terms: conditions — Pulmonary Atelectasis; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional (Active Comparator)
  Interventions: Procedure: conventional recruitment maneuvers
- ultrasound-guided (Active Comparator)
  Interventions: Procedure: ultrasound-guided recruitment maneuvers

INTERVENTIONS:
Procedure: conventional recruitment maneuvers — The recruitment maneuver will be performed at 3 predefined time points: 5 minutes after induction of GA (T2), 5 minutes after insufflation of the capnoperitoneum (T3), After the end of surgery and before recovery from anesthesia (T4).
  by pressure controlled mode starting with an airway pressure of 15 cmH2O the subsquently changed ( decrease or increase) to provide targeted tidal volume according to each patient, maintaining end-tidal carbon dioxide between 35 to 45 mmHg with 5 cmH2O increments in PEEP until a peak pressure of 30 cmH2O will be achieved. Each PEEP level will be maintained for 5 s. The peak airway pressure will be maintained for 10 s or five breaths and subsequently reduced, followed by maintenance with the previous ventilator settings
  Other Names: control
  Arms: conventional
Procedure: ultrasound-guided recruitment maneuvers — * Ultrasound guided maneuver will be performed at T2, T3 and T4.
  * The recruitment maneuver will be performed under ultrasound guidance until no collapsed lung area is visible. The strategy to increase the airway pressure will be the same as that for the conventional maneuver, although the maximal pressure limit will be 40 cmH2O. The Recruitment maneuvers (RM) will be started searching the pressure level at which the consolidation pattern disappears and progressive lung re-aeration is observed and will be recorded for all patients (the lung's opening pressure).(14) Lung ultrasound examination will be performed every 5 cmH2O increments in PEEP to detect the lung's opening pressure.
  Arms: ultrasound-guided

SUMMARY:
In anesthetized children, the incidence of lung collapse with episodes of hypoxemia is high. Diaphragmatic dysfunction induced by general anesthesia is one of the most important factors in the genesis of regional losses of lung aeration. The mass of the abdominal organs pushes the diaphragm cranially compressing the lungs in the most dependent areas. Such regional lung collapse may range from a slight loss of aeration to complete atelectasis.

DETAILED DESCRIPTION:
A wide variety of recruitment maneuvers has been described. The most relevant are represented by sustained inflation maneuvers, high pressure-controlled ventilation, incremental PEEP, and intermittent sighs. However, the best recruitment maneuver technique is currently unknown and may vary according to the specific circumstances. The most commonly used recruitment maneuver is the sustained inflation technique, in which a continuous pressure of 40 cm H2O is applied to the airways for up to 60 seconds. Sustained inflation has been shown to be effective in reducing lung atelectasis, improving oxygenation and respiratory mechanics, and preventing endotracheal suctioning-induced alveolar derecruitment. However, the efficacy of sustained inflation has been questioned and other studies showed that this intervention may be ineffective, short-lived, or associated with circulatory impairment, an increased risk of baro/volutrauma, a reduced net alveolar fluid clearance, or even worsened oxygenation.

Lung ultrasound has been gaining consensus as a noninvasive, radiation-free tool for diagnosing various pulmonary diseases in adult and pediatric patients. Evidence supporting lung ultrasound use is expanding beyond emergency and critical care settings to perioperative care.

It has been reported that lung ultrasound (LUS) at a patient's bedside immediately following surgery can be useful for diagnosing respiratory complications. LUS has been proven to be a valuable bedside diagnostic tool for pneumothorax, with high sensitivity and specificity (78.6% and 98.4%, respectively), and a higher rate of detecting abnormalities such as lung alveolar consolidation and pleural effusion than bedside chest X-ray or physical examination. LUS has also been used to diagnose anesthesia-induced atelectasis in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic abdominal surgery
* American Society of anaesthesiologist class I & II

Exclusion Criteria:

* Pre-existing cardiac disease.
* Morbidly obese patients according to age.
* Patients with previous thoracic or cardiac surgery.
* Upper or lower airway infection within 2 weeks before the surgery.
* Lung ultrasound abnormalities including patches, pneumothorax, and pleural effusion.
* Abnormal preoperative chest x-ray findings including atelectasis, pneumothorax, pleural effusion or pneumonia.
* Preoperative oxygen saturation measured by pulse oximetry (SpO2) of 96% or less on room air.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The incidence of atelectasis | postoperative first 2 hours
  The incidence of atelectasis in post anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: hoda ezz, Principal Investigator — tanta university, faculty of medicine
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No